CLINICAL TRIAL: NCT05750524
Title: The Effect of Hand Massage Applied With Two Different Methods on Endotracheal Suctioning Pain and Hemodynamic Parameters
Brief Title: The Effect of Hand Massage on Endotracheal Suctioning Pain and Hemodynamic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ilkin Yilmaz, Assist Prof., Ph.D., Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 7074-GOA
Record Dates: First submitted 2023-02-03; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Endotracheal Aspiration; Pain; Reflexology; Massage; Hemodynamic Instability
Keywords: endotracheal suctioning; endotracheal aspiration; pain; hand massage; reflexology; hemodynamic parameters
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: In the AB trial group, reflexology hand massage will be applied on the first day, classical hand massage on the second day, and in the BA group classical hand massage on the first day and reflexology hand massage on the second day will be applied.
Who Masked: Participant, Investigator
Masking Description: Patients and the investigator doing the suctioning and assessing the patient's pain and vital signs will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reflexology (Experimental): In the reflexology group, reflexology hand massage applied between two suctioning period
  Interventions: Other: reflexology hand massage
- classical massage (Placebo Comparator): In the classical massage group, classical hand massage applied between two suctioning period
  Interventions: Other: classical hand massage

INTERVENTIONS:
Other: reflexology hand massage — Reflexology massage methods applied randomly to both trial groups.
  Arms: reflexology
Other: classical hand massage — Classical hand massage methods applied randomly to both trial groups.
  Arms: classical massage

SUMMARY:
Endotracheal suctioning (ETS) is one of the most frequently applied care procedures in intensive care units in patients with artificial airway and mechanical ventilation. Suctioning, like all other invasive procedures, causes some complications. Various complications such as pain, hypoxemia, irregularity in blood pressure and heart rate, arrhythmia, increased respiratory frequency, and decreased respiratory depth may develop in patients. Pain is a physiological response that affects the patient's comfort and vital signs. hemodynamic parameters triggered by suctioning, as well as pain, may be positively affected by reflexology and classical hand massage.

DETAILED DESCRIPTION:
Endotracheal suctioning (ETS) is one of the most frequently applied care procedures in intensive care units in patients with artificial airway and mechanical ventilation. ETS is applied to patients for purposes such as ensuring airway opening in patients by removing secretions from the lungs, ensuring and maintaining optimal gas exchange.

Suctioning, like all other invasive procedures, causes some complications. Various complications such as pain, hypoxemia, irregularity in blood pressure and heart rate, arrhythmia, increased respiratory frequency, and decreased respiratory depth may develop in patients. In the literature, endotracheal suctioning has been reported as one of the most painful procedures reported by patients in the intensive care unit, regardless of the application technique. Pain is a physiological response that affects the patient's comfort and vital signs. In the literature, there are studies on music therapy to reduce or completely relieve the pain related to the suctioning procedure, but there are no studies applied with other alternative methods.

Classical hand massage and reflexology hand massage are included in complementary and supportive applications. It is stated that reflexology massage applied in studies on various patient groups is effective on many symptoms such as fatigue, pain, anxiety, sleep and cramps. There was no study finding that examined the effect of hand massage on suctioning pain and hemodynamic parameters during suctioning. It is thought that hand massage can be an effective intervention that nurses can apply independently in the management of pain during suctioning. It is thought that hemodynamic parameters triggered by suctioning, as well as pain, will be positively affected by reflexology and classical hand massage.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Those who agreed to participate in the study
* Orally intubated,
* Receiving mechanical ventilator support,
* No history of chronic pain (eg arthritis)
* Not addicted to alcohol and drugs
* Does not have a psychological problem (such as depression, anxiety disorder),
* Not using anxiolytic, antidepressant or antipsychotic medication
* The sedation-analgesic levels did not change during the study,
* No additional sedation-analgesic medication is applied during the massage and suctioning applications,
* Riker Sedation Agitation Scale score is 2-4 points,
* Having no objections to massaging their hands (not having any skin lesions, burns, pathological diseases related to muscles and bones),
* Patients who need suctioning within two hours at the latest after the end of the massage will be included in the sample.

Exclusion Criteria:

* Being under the age of 18,
* Having a Riker Sedation Agitation Scale score of 1, or 5 and above,
* Changing sedation and analgesic doses during the study,
* Having chronic disease pain,
* Being addicted to alcohol and drugs,
* Having a psychological problem and using antidepressant, anxiolytic or antipsychotic medication,
* Discharged, exitus, extubated, tracheostomy or tracheostomy opened,
* Having any skin lesions, burns, open wounds, pathological diseases related to muscles and bones on their hands,
* Needing suctioning during the massage application,
* Not needing suctioning within the first two hours after the massage application is finished,
* Patients who require suctioning within one hour after the first suctioning procedure performed between 08:00-20:00 will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
change from baseline pain level of patients at 5 minutes both reflexology and classical hand massage group | just before ETS and immediately after and 5th minute after ETS
  pain level (point) was measured via Critical-care Pain Observation Tool just before ETS and immediately after and 5th minute after ETS before and after massages

SECONDARY OUTCOMES:
blood pressures of patients both reflexology and classical hand massage group | just before ETS and immediately after and 5th minute after ETS
  systolic and diastolic blood pressure (mmHg) were measured just before ETS and immediately after and 5th minute after ETS before and after massages
heart rate of patients both reflexology and classical hand massage group | just before ETS and immediately after and 5th minute after ETS
  heart rate (heart rate/minute) was measured just before ETS and immediately after and 5th minute after ETS before and after massages
respiratory frequency of patients both reflexology and classical hand massage group | just before ETS and immediately after and 5th minute after ETS
  respiratory frequency (respiratory frequency/minute) measured just before ETS and immediately after and 5th minute after ETS before and after massages
tidal volume of patients both reflexology and classical hand massage group | just before ETS and immediately after and 5th minute after ETS
  tidal volume (ml) was measured just before ETS and immediately after and 5th minute after ETS before and after massages
peripheral oxygen saturation of patients both reflexology and classical hand massage group | just before ETS and immediately after and 5th minute after ETS
  peripheral oxygen saturation (%) measured just before ETS and immediately after and 5th minute after ETS before and after massages

CONTACTS AND LOCATIONS:
Overall Officials: İlkin Yılmaz, PhD, Study Chair — Assist Prof; Gizem Göktuna, PhDc, Principal Investigator — Res Assis; Gülşah Gürol Arslan, PhD, Principal Investigator — Assoc Prof; Dilek Özden, PhD, Principal Investigator — Professor
Locations (1):
- Ilkin Yilmaz, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We cannot share participant data due to Turkish Personal Data Protection Law no. 6698

REFERENCES:
- See also: Yaman Aktaş, Y., & Karabulut, N. (2016). The effects of music therapy in endotracheal suctioning of mechanically ventilated patients. Nursing in Critical Care, 21(1), 44-52. — https://pubmed.ncbi.nlm.nih.gov/25721305/
- See also: Acikgoz, A., & Yildiz, S. (2015). Effects of Open and Closed Suctioning Systems on Pain in Newborns Treated with Mechanical Ventilation. Immunology and Allergy Clinics of North America, 35(4), 653-663. — https://doi.org/10.1016/j.pmn.2015.01.002
- See also: Wang, H. L., & Keck, J. F. (2004). Foot and hand massage as an intervention for postoperative pain. Pain Management Nursing, 5(2), 59-65. — https://doi.org/10.1016/j.pmn.2004.01.002
- See also: Özden, D., & Görgülü, R. S. (2015). Effects of open and closed suction systems on the haemodynamic parameters in cardiac surgery patients. Nursing in Critical Care, 20(3), 118-125. — https://pubmed.ncbi.nlm.nih.gov/24991700/